CLINICAL TRIAL: NCT06312007
Title: Semi-seated Holding Position to Reduce Stress Responses in Spontaneous Crying Newborn in the Neonatal Intensive Care Unit
Brief Title: Semi-seated Holding Position to Reduce Stress Responses in in the Neonatal Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Andi Dwi Bahagia Febriani, dr, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UH23030202
Record Dates: First submitted 2024-02-29; First posted 2024-03-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Semi Seated Position; Side Lying Position
Keywords: semi seated position, cortisol saliva, oxytocin saliva
MeSH Terms: interventions — Facilitated Tucking

STUDY DESIGN:
Intervention Model Description: Intervention semi seated position Control side lying position
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi-seated position (Experimental): Semi seated position
  Interventions: Other: Semi seated position; Other: side lying position
- Side Lying position (Experimental): Side lying position
  Interventions: Other: Semi seated position; Other: side lying position

INTERVENTIONS:
Other: Semi seated position — The patient is positioned 45-90 degrees
  Other Names: Half sitting position
Other: side lying position — Side lying position
  Other Names: facilitated tucking

SUMMARY:
This study to compare half semi seated position and side lying position with cortisol level on the neonate's stress respon

DETAILED DESCRIPTION:
This study was a randomized control trial with inclusion criteria of moderately preterm, late preterm, and term baby. Exclusion criteria were babies experiencing respiratory distress and multiple congenital anomalies. Two treatments were carried out, the first was in a semi-seated position, the second was the control group, given the side lying position, then the levels of cortisol and salivary oxytocin were compared to see the stress response.

ELIGIBILITY:
Inclusion Criteria:

* Modertely preterm, late preterm, aterm

Exclusion Criteria:

* neonates with respiratory distress
* multiple congenital anomali

Ages: 32 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Kortisol level | 20 weeks
  Level of cortisol after semi seated and side lying position
Oxytocin level | 20 weeks
  Level of oxytocin saliva after semi seated and side lying position

CONTACTS AND LOCATIONS:
Locations (1):
- Hasanuddin University, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Other researchers can contact us via email if they want to know about our research
Supporting Information: Study Protocol, SAP
Time Frame: 2024-2025